CLINICAL TRIAL: NCT07106918
Title: A Randomized, Double-blind, Placebo/Positive Control Phase Ia Clinical Trial Evaluating the Safety, Tolerability, and Pharmacokinetics of SIBP-A16 Injection in Healthy Adults
Brief Title: A Clinical Trial of SIBP-A16 Injection in Healthy Adults
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Shanghai Institute Of Biological Products (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: SIBP-A16-I
Record Dates: First submitted 2025-07-30; First posted 2025-08-06 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-07

CONDITIONS: Respiratory Syncytial Virus (RSV)
Keywords: Respiratory syncytial virus; SIBP-A16; safety; tolerability; pharmacokinetics
MeSH Terms: interventions — nirsevimab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- SIBP-A16 injection (Experimental): Strength: dose 1, dose 2 dose 3 and dose 4. The participants enrolled will be randomly assigned to different dose groups, and they will be enrolled in groups according to the dose from low to high.
  Interventions: Biological: SIBP-A16 injection
- Nirsevimab (Active Comparator): Participants injected Nirsevimab will compare with participants in dose 2 experimental group.
  Interventions: Biological: Nirsevimab
- SIBP-A16 buffer solution (Placebo Comparator): Participants in the placebo group from different queues will receive the same dose as the corresponding experimental group
  Interventions: Other: SIBP-A16 buffer solution

INTERVENTIONS:
Biological: SIBP-A16 injection — Single administration via intramuscular or intravenous injection. All participants received a single injection of the corresponding dose.
  Arms: SIBP-A16 injection
Biological: Nirsevimab — Single administration via intramuscular.
  Arms: Nirsevimab
Other: SIBP-A16 buffer solution — Single administration via intramuscular or intravenous injection. All participants received a single injection of the corresponding dose.
  Arms: SIBP-A16 buffer solution

SUMMARY:
This study is a randomized, double-blind, placebo/positive control Phase Ia clinical trial evaluating the safety, tolerability, and pharmacokinetics of SIBP-A16 injection in healthy adults

DETAILED DESCRIPTION:
This study plans to set up 5 queues, with queues 1, 3, 4, and 5 each containing 20 participants in the experimental group and 4 participants in the placebo group. Queue 2 contains 20 participants in the experimental group, 20 participants in the positive control group, and 4 participants in the placebo group. The total number of participants included in the five queues is 140. SIBP-A16 injection and placebo will be administered in four different doses and two different ways of administration. The study adopted a sequential injection design. After completing a 14-day preliminary safety observation of drug administration in the previous group, the Safety Review Committee (SRC) will conduct a preliminary safety assessment. Once the SRC evaluation results are safe (not meeting the dose escalation termination criteria), the next group will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals aged 18 to 45 on the day of enrollment, regardless of gender.
* Male body weight ≥ 50.0 kg, female body weight ≥ 45.0 kg, BMI between 19.0 and 27.0 kg/m2 (including critical values).
* Screening period physical examination, vital sign examination, 12 lead electrocardiogram, chest X-ray or clinical laboratory examination, and other auxiliary examination results show normal or abnormal without clinical significance as judged by the researcher.
* Individuals who voluntarily participate in clinical trials and sign informed consent forms.
* Individuals are able to communicate well with the researchers and understand and comply with the requirements of this study.

Exclusion Criteria:

* Known to have a history of serious clinical diseases such as mental system, circulatory system, endocrine system, digestive system, respiratory system, hematological and metabolic abnormalities, or any other diseases that can interfere with the test results.
* Individuals with a history of drug allergies or specific allergies, or individuals with allergies, or those known to be allergic to the components or analogues of this drug.
* During the screening period, individuals with abnormal results from physical examination, laboratory tests and clinical significance were identified by the researchers as having an impact on the evaluation of this trial.
* During the screening period, male individuals with QTcF ≥ 450 milliseconds and female individuals with QTcF ≥ 470 milliseconds on electrocardiogram.
* Individuals who have received monoclonal/polyclonal antibody drugs within 6 months prior to screening.
* Individuals have received immunoglobulin or blood product treatment within 6 months prior to screening.
* Individuals who have received passive immune agents, immunosuppressants, or corticosteroids within the 6 months prior to screening.
* Individuals who experience acute illnesses such as fever ≥ 37.3 ℃ (armpit temperature) and diarrhea within one week before their first medication.
* Individuals experienced symptoms and signs of acute upper respiratory tract infection within 2 weeks prior to the first use of medication.
* Individuals who have received the respiratory syncytial virus (RSV) vaccine in the past.
* Individuals have received any vaccine within 30 days prior to screening.
* Select individuals who have smoked at least 5 cigarettes per day within the first 3 months and those who cannot quit smoking throughout the entire trial period.
* Individuals with an average weekly alcohol consumption of ≥ 14 units within the first 3 months of screening, or those who cannot abstain from alcohol during the trial period.
* Individuals have a history of long-term excessive consumption of tea, coffee, or caffeinated beverages.
* Individuals have used any medication or health supplement within the 14 days prior to screening.
* Individuals with a history of drug abuse/dependence or drug use within the past year prior to screening.
* Screening individuals who have participated in any drug clinical trials and have used the investigational drug within the previous 3 months.
* Individuals with a history of blood donation or significant bleeding within the previous 4 weeks prior to screening, or those planning to donate blood or blood components during the study period.
* Pregnant or lactating women.
* Those who have plans to conceive, donate sperm or eggs, or are unable to voluntarily take effective contraceptive measures during the trial period (including partners).
* Those who have special dietary requirements and cannot follow a reasonable and normal diet.
* The researchers believe that the individuals may have other situations that may affect compliance or be unsuitable to participate in this trial

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 140 (Estimated)
Dates: Start 2025-08-17 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
AE (Adverse Events) | From day 1 to day 361 after administration
  That is adverse events, any adverse events that occurred to the participant during the study period.
SAE (Serious Adverse Events) | From day 1 to day 361 after administration
  That is serious adverse events, any serious adverse events that occurred to the participant during the study period.
Adverse Event of Special Interest (AESI) | From day 1 to day 361 after administration
  Adverse events defined in the protocol that require special attention, such as abnormal liver function, etc.

SECONDARY OUTCOMES:
AUC (Area Under The Plasma Concentration Versus Time Curve) | Based on multiple pharmacokinetic blood collection points specified in the protocol
  It shows the degree to which a drug is absorbed and used in the body.
Cmax (Peak Plasma Concentration) | Based on multiple pharmacokinetic blood collection points specified in the protocol
  It shows the highest plasma concentration of a drug that can be achieved after administration.
Tmax (Peak Time) | Based on multiple pharmacokinetic blood collection points specified in the protocol
  That is peak time of drug action, it shows the time required to reach the maximum concentration on the participant plasma concentration curve after administration.

OTHER OUTCOMES:
Level of Anti-drug antibody (ADA) | Before injection, on the 15th, 31st, 91st, 151st, 271st, and 361st days after administration
  If ADA is positive, further check the levels of neutralizing antibodies against SIBP-A16 or neutralizing antibodies against Nisevere monoclonal antibody

CONTACTS AND LOCATIONS:
Overall Officials: Chao lin Huang, Principal Investigator — Wuhan Jinyintan Hospital
Locations (1):
- Wuhan Jinyintan Hospital, Wuhan, China

IPD SHARING:
Plan to Share IPD: No